CLINICAL TRIAL: NCT01743612
Title: Laser SPEckle Contrast Imaging Interest in dEtection of Cutaneous Microvascular Dysfunction in Systemic Sclerosis.
Brief Title: Laser Speckle Contrast Imaging for Cutaneous Microvascular Dysfunction Detection in Systemic Sclerosis.
Acronym: SPECIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DCIC 11 25
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2015-12

CONDITIONS: Raynaud Disease; Scleroderma, Systemic
Keywords: healthy subject; hand blood flow; laser speckle contrast imaging
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic | interventions — Laser Speckle Contrast Imaging; Cool-Down Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sclerodermic patients (Experimental): patients with systemic sclerosis according to Leroy's classification
  Interventions: Procedure: laser speckle contrast imaging; Procedure: Cooling
- Primary Raynaud's phenomenon (Experimental): without secondary disease
  Interventions: Procedure: laser speckle contrast imaging; Procedure: Cooling
- Healthy subjects (Experimental): 18 years old or more
  Interventions: Procedure: laser speckle contrast imaging; Procedure: Cooling

INTERVENTIONS:
Procedure: laser speckle contrast imaging — blood flow recording during 30 minutes after 2 post-occlusive hyperaemia of 5 minutes separated by 30 minutes.
Procedure: Cooling — blood flow of the hand recording during 30 minutes in a cooling-box

SUMMARY:
The aim of the study is to determine if postocclusive hyperemia of palmar and dorsal face of the hand with Laser speckle contrast imaging discriminate between patients with systemic sclerosis, subjects with primary Raynaud's phenomenon and healthy subjects.

DETAILED DESCRIPTION:
Microvascular dysfunction is a key event in the pathogenesis of systemic sclerosis. There are currently no test measuring it in clinical practice. Response to humeral occlusion is interesting and this response has been studied with laser Doppler flowmetry. More recently, laser imaging has been used analysing the granularity of the laser: laser Speckle Contrast Imaging which allow combining high temporal resolution to high spatial resolution.

The investigators proposed, in this study, to compare this imaging at basal and after post-occlusive hyperaemia of dorsal and palmar face of hand in 3 groups: healthy subjects, primary Raynaud's phenomenon and systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects:
* Man ou woman 18 years old or more.
* Without Raynaud's phenomenon or systemic sclerosis.

Raynaud's phenomenon subjects:

* Man ou woman 18 years old or more.
* with primary Raynaud's phenomenon.

Systemic sclerosis:

* Man ou woman 18 years old or more.
* systemic sclerosis in accordance to Leroy's classification.

Exclusion Criteria:

* active digital ulceration
* Bosentan, iloprost ou sildenafil treatment
* History of axillary dissection , trauma or surgery
* history of thromboembolic disease or thrombophilia
* minor or law-protected major
* exclusion period in another study
* No affiliation to medicare
* pregnant, parturient or breasting woman
* concomitant serious disease: progressive cancer, liver failure, history of myocardial infarction less than 5 years, angor
* smoking in the 6 last months
* person deprived of liberty by a legal or administrative decision, person under legal protection
* maximal annual indemnification reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Post-occlusive hyperemia response between groups | 30 minutes
  The range of post-occlusive hyperemia response will be compared between the 3 arms.

SECONDARY OUTCOMES:
post-occlusive hyperemia response between zones | 30 minutes
  The range of post-occlusive hyperemia response will be compared between zones.
abnormal post-occlusive hyperemia response and finger pad scars | 30 minutes
  comparison of range of post-occlusive hyperemia response with or without finger pad scars.
Entropy and Fourier transform | 30 minutes
  The interest of the signal analyses to distinguish systemic sclerosis, raynaud's phenomenon and healthy subjects will be studied with entropy and Fourier transform.
Post-occlusive hyperemia response between the 2 faces | 30 minutes
  The Range of post-occlusive hyperemia response will be compared between the 2 hand faces (palmar and dorsal).

OTHER OUTCOMES:
Blood flow after cooling between groups | 30 minutes
  Range of the diminution of blood flow in palmar and dorsal hand faces will be compared in the 3 groups
reproductibility of hand cooling | Day 0 and Day 4
  The reproductibility of the measure of blood flow after cooling will be studied twice, at day0 and 4 days later.
blood flow after cooling in each group | 30 minutes
  The range of blood flow after cooling on pulpar and dorsal face of hand will be compared between the 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD, PhD, Principal Investigator — CIC, CHU Grenoble
Locations (2):
- France (2):
  - Clinical Research Center, Grenoble
  - Vascular Medical Unit, Grenoble

REFERENCES:
- [Derived] Gaillard-Bigot F, Roustit M, Blaise S, Gabin M, Cracowski C, Seinturier C, Imbert B, Carpentier P, Cracowski JL. Abnormal amplitude and kinetics of digital postocclusive reactive hyperemia in systemic sclerosis. Microvasc Res. 2014 Jul;94:90-5. doi: 10.1016/j.mvr.2014.05.007. Epub 2014 Jun 2. PMID 24990822